CLINICAL TRIAL: NCT07373665
Title: Enhancing Critical Thinking, Clinical Decision-Making, and Knowledge Retention Utilizing Problem-Based Learning: A Cluster Randomized Controlled Trial Among Obstetric Nursing Students
Brief Title: Problem-Based Learning to Improve Critical Thinking in Obstetric Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eman Atef Elsokary (Other)
Collaborators: Helwan University (Other)
Responsible Party: Sponsor-Investigator, Eman Atef Elsokary, Lecturer of Maternal and Newborn Health Nursing, Benha University
Organization: Benha University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PBL-OBN-2025
Record Dates: First submitted 2026-01-21; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Problem-based Learning in Nursing Education
Keywords: Problem-based learning; Nursing education; Obstetric nursing; Critical thinking; Clinical decision making; Knowledge retention; Undergraduate nursing students; Educational intervention; Cluster randomized trial

STUDY DESIGN:
Intervention Model Description: Participants were assigned to intervention or control groups using cluster randomization at the academic-group level to minimize contamination. Academic clusters were allocated in parallel to either problem-based learning (PBL) or traditional lecture-based instruction. All clusters were followed concurrently, and outcomes were assessed at baseline, immediately post-intervention, and at four-week follow-up.
Masking Description: This was an open-label educational intervention. Due to the nature of the instructional methods, participants, instructors, and investigators were aware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem-Based Learning (PBL) Group (Experimental): Participants in this arm received a structured problem-based learning (PBL) instructional program covering normal labor, preeclampsia/eclampsia, and postpartum hemorrhage. The intervention was delivered in small-group sessions using standardized clinical case scenarios, guided facilitation, self-directed learning, and group discussion over a six-week period.
  Interventions: Behavioral: Problem-Based Learning (PBL)
- Traditional Lecture-Based Instruction Group (Active Comparator): Participants in this arm received traditional lecture-based instruction covering normal labor, preeclampsia/eclampsia, and postpartum hemorrhage, delivered through instructor-led lectures and PowerPoint presentations in accordance with the standard course syllabus.
  Interventions: Behavioral: Traditional Lecture-Based Instruction

INTERVENTIONS:
Behavioral: Problem-Based Learning (PBL) — A structured problem-based learning instructional approach using standardized clinical case scenarios related to maternal and newborn health nursing. The intervention emphasized active learning, small-group discussion, self-directed learning, clinical reasoning, and facilitated synthesis of evidence-based nursing decisions.
  Arm Assigned:Problem-Based Learning (PBL) Group
  Arms: Problem-Based Learning (PBL) Group
Behavioral: Traditional Lecture-Based Instruction — Traditional lecture-based instruction delivered through instructor-led teaching and PowerPoint presentations, covering maternal and newborn health nursing topics according to the standard undergraduate nursing curriculum.
  Arm Assigned:Traditional Lecture-Based Instruction Group
  Arms: Traditional Lecture-Based Instruction Group

SUMMARY:
This study examined the effect of a problem-based learning (PBL) instructional approach on undergraduate nursing students' learning outcomes in obstetrics health nursing. The intervention was implemented with nursing students at the Faculty of Nursing, Benha University, Egypt.

Students participated in structured problem-based learning sessions designed to enhance critical thinking, clinical decision making, and knowledge retention related to maternal and newborn health topics. Learning outcomes were assessed before and after the intervention using validated assessment tools.

The findings of this study aim to provide evidence on the effectiveness of problem-based learning as an educational strategy in nursing education and to inform curriculum development and teaching practices in obstetrics health nursing Course.

DETAILED DESCRIPTION:
This study is a cluster randomized controlled trial designed to evaluate the effect of a problem-based learning (PBL) instructional approach on critical thinking, clinical decision-making, and knowledge acquisition and retention among undergraduate obstetric nursing students. The study was conducted in classroom settings at the Faculty of Nursing, Benha University, Benha, Egypt, during the first semester of the 2025-2026 academic year.

Eligible participants were third-level undergraduate nursing students enrolled in the obstetrics nursing course. Academic groups were used as the unit of randomization to minimize contamination between students. From the available academic groups, 12 clusters were randomly selected and allocated in a 1:1 ratio to either the intervention group (PBL) or the control group (traditional lecture-based instruction). All eligible students within the selected clusters were included, resulting in a total sample of 312 students.

At baseline, participants in both groups completed assessments measuring demographic characteristics, knowledge acquisition, critical thinking, and clinical decision-making. Following baseline assessment, control clusters received traditional lecture-based instruction covering normal labor, preeclampsia/eclampsia, and postpartum hemorrhage according to the standard course syllabus. Intervention clusters participated in a structured PBL program addressing the same topics using standardized clinical case scenarios and guided facilitation. The intervention emphasized problem identification, self-directed learning, group discussion, and application of knowledge to clinical decision-making.

Outcome measures were collected immediately after completion of the instructional period and again four weeks later to evaluate knowledge retention and sustained development of critical thinking and clinical decision-making skills. Validated instruments were used to assess critical thinking and clinical decision-making, while a researcher-developed, case-based multiple-choice questionnaire was used to assess knowledge acquisition and retention. Ethical approval was obtained from the Scientific Research Ethics Committee of the Faculty of Nursing, Helwan University prior to study initiation. Participation was voluntary, and informed consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Undergraduate nursing students enrolled in the third academic level of the Obstetrics and Gynecology Nursing course at the Faculty of Nursing, Benha University.
2. Aged 18 to 21 years at the time of enrollment.
3. Regular attendance in the course during the study period.
4. Willingness to participate and provide written informed consent.
5. No prior formal exposure to structured problem-based learning (PBL).
6. Completion of baseline assessment prior to participation.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 312 (Actual)
Dates: Start 2025-09-20 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Critical Thinking Skills | Baseline (pre-intervention), immediately post-intervention, and 4-week follow-up
  Critical thinking skills were assessed using the Critical Thinking Questionnaire (CThQ), a validated 25-item self-administered instrument measuring six domains of critical thinking: remembering, understanding, applying, analyzing, evaluating, and creating. Items are rated on a 5-point Likert scale, with higher scores indicating stronger critical thinking ability.
Clinical Decision-Making Ability | Baseline (pre-intervention), immediately post-intervention, and 4-week follow-up
  Clinical decision-making ability was measured using the Clinical Decision Making in Nursing Scale (CDMNS), a validated 40-item self-report instrument assessing four dimensions of decision-making: search for alternatives, canvassing of objectives and values, evaluation of consequences, and information search. Higher total scores reflect more developed clinical decision-making abilities.
Knowledge retention in obstetrics Health Nursing | Baseline (pre-intervention), immediately post-intervention, and 4-week follow-up
  Knowledge acquisition and retention were assessed using a researcher-developed, case-based multiple-choice questionnaire covering normal labor, preeclampsia/eclampsia, and postpartum hemorrhage. The tool consists of 30 items, with higher scores indicating higher levels of knowledge acquisition and retention.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Atef Elsokary, PhD, Principal Investigator — Faculty of Nursing, Helwan University, Egypt
Locations (1):
- Faculty of Nursing, Benha University, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No